CLINICAL TRIAL: NCT02858531
Title: Predictive Tracking of Patient Flow in the Emergency Services During the Virus Winter Epidemics
Acronym: PREDAFLU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1508191; 1969303 v 0 (Other: CNIL)
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Disease Outbreaks; Child; Elderly; Bronchiolitis; Acute Renal Failure
MeSH Terms: conditions — Bronchiolitis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients < 24 months or 60 years with bronchiolitis or ARF: ARF = Acute Renal Failure
  Interventions: Other: data retrieval

INTERVENTIONS:
Other: data retrieval — data retrieval with the Hospital Information System

SUMMARY:
Epidemics and infectious diseases in general, punctuate much of the activity of an emergency service. The impact of winter infections is particularly important to vulnerable populations such as infant during bronchiolitis epidemics and the elderly during seasonal influenza. Each year, these epidemic phenomena lead to disorganization of emergency services and healthcare teams by lack of anticipation and organizational measures in particular to manage the approval of emergency services for the most vulnerable populations requiring hospitalization.

For 2 years, the pediatric emergency department of St Etienne University Hospital has a decision support tool for the periods of winter epidemics. Through a retrospective analysis of Passages of Emergency summary, this tool provides an estimate of infants with bronchiolitis flow day to day, and the availability in real time of an abnormally high flow of patients to pediatric emergencies. These data can help to affirm that the epidemic begins in this hospital.

ELIGIBILITY:
Inclusion Criteria:

* child < 24 months with bronchiolitis
* elderly < 60 years with acute renal failure or breathing problem

Exclusion Criteria:

* refuse of transmission of their data

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: child < 24 months with bronchiolitis or elderly < 60 years with acute renal failure
Sampling Method: Non-Probability Sample
Enrollment: 760000 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
build a predictive tool | at inclusion
  a tool with different levels of alerts of the influx of people aged to emergencies during winter epidemics.
  Variables in the model : activity database in emergency services, computer data, virology database and average length of stay.

SECONDARY OUTCOMES:
Difference between the estimated date and the effective date of the activity peak on the average length of stay of patients in the hospital of Saint Etienne | at inclusion
Difference between the estimated date and the effective date of the activity peak on the average length of stay of patients in the other hospitals | at inclusion
Comparison virological databases with clinical diagnosis of patients | at inclusion
Percentage of elderly staying more than 10 hours in the emergency services. | at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MORY, MD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (11):
- France (11):
  - CHU de Grenoble (adult emergency service), Grenoble
  - CHU de Grenoble (pediatric service), Grenoble
  - CHU de Lyon (adult emergency service), Lyon
  - CHU de Lyon (laboratory of virology), Lyon
  - CHU de Lyon HFME (pediatric service), Lyon
  - CHU de Saint Etienne (adult emergency service), Saint-Etienne
  - CHU de Saint Etienne (Pediatric service), Saint-Etienne
  - CH de Valence (adult emergency service), Valence
  - CH de Valence (pediatric service), Valence
  - CH de Villefranche (adult emergency service), Villefranche-sur-Saône
  - CH de Villefranche (pediatric service), Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No